CLINICAL TRIAL: NCT05205733
Title: Expanding Fertility Care to Poor and Low Resourced Settings Study
Acronym: EXPLORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-33495
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy; Male Infertility; Infertility, Male; Fertility Disorders
Keywords: Disparities; Resource limited; Low-resource communities
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Participants are assigned to complete either a mail-in or in-clinic semen analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Clinic Semen Analysis Testing (No Intervention): Men needing semen analysis for infertility work-up.
- No in-clinic semen analysis testing (Experimental): Men needing semen analysis for infertility work-up.
  Interventions: Other: Mail-in semen analysis kit

INTERVENTIONS:
Other: Mail-in semen analysis kit — Presumably an easier, convenient, and more comfortable way to provide a semen analysis with an in-home mail-in semen analysis kit
  Other Names: Fellow Health Semen Analysis
  Arms: No in-clinic semen analysis testing

SUMMARY:
The investigators currently lack an understanding of barriers to completing the male factor infertility evaluation. Furthermore, as the investigators continue to expand access to fertility treatment particularly within low-resourced settings, it is important that all aspects of infertility within a couple are equally explored. The COVID-19 pandemic has disproportionately affected low-income communities and communities of color at greater rates in terms of not only disease morbidity/mortality but how medical systems are accessed and care is delivered.

DETAILED DESCRIPTION:
This pilot study was designed to help providers identify barriers to completing the basic infertility work-up in a low resource setting with a focus on accessibility and feasibility of semen analysis testing. As a pilot study, a total of 60 male partners of patients who are seeking infertility treatment at the Zuckerberg San Francisco General Hospital Gynecology clinic will be recruited. Participants will be randomized to completing a semen analysis by either the standard in-clinic test or an at-home sperm testing kit. The investigators hypothesis is that there will be an increase in participants completing their semen analysis when using the at-home sperm testing kit as opposed to having to come to the lab.

Specific Aims:

1. To identify barriers to completing a semen analysis.
2. To compare barriers unique to completing an in-clinic versus at-home testing.
3. To compare satisfaction scores with in-clinic versus at-home testing.
4. To compare the time to complete the semen analysis with in-clinic versus at-home testing.
5. To compare the time to initiating treatment after completing in-clinic versus at-home testing.

Patients seen at Zuckerberg San Francisco General who are currently undergoing an infertility evaluation as a part of the basic infertility assessment will be contacted. Consented participants will be randomized to complete an at home vs. lab semen analysis. After the semen analysis is completed, participants will be sent a comprehensive questionnaire regarding their experience, level of satisfaction, and barriers with completion of the recent semen analysis. Participants will be given 3 months to complete the semen analysis. If not completed in this timeframe, participants will be sent a different comprehensive questionnaire regarding their barriers with completion of the semen analysis. Additional clinical questions include time from semen analysis order to completion as well as time from semen analysis completion to start of treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* All English or Spanish speaking male partners of female patients undergoing an infertility work-up evaluation at Zuckerberg San Francisco General Hospital and recommended to undergo a semen analysis as a part of this workup.

Exclusion Criteria:

* If they do not speak English or Spanish they will be excluded
* If they are under the age of 18 y.o
* If they are not recommended to undergo a semen analysis as a part of the infertility evaluation
* If they are unable to produce a semen sample.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To compare the time to complete the semen analysis with in-clinic versus at-home testing. | 3 months after consented to the study.
  The time to completion between in-clinic versus at-home testing will be identified when the provider obtains the results.

SECONDARY OUTCOMES:
To identify barriers to completing a semen analysis. | Three months after being consented to the study.
  The barriers will be identified via a survey to be completed by the participant.
To compare barriers unique to completing an in-clinic versus at-home testing. | Three months after being consented to the study.
  The unique barriers will be identified via a survey to be completed by the participant.
To compare satisfaction scores with in-clinic versus at-home testing. | Three months after being consented to the study.
  Patient satisfaction will be identified via a survey using the Likert Scale to be completed by the participant where strongly agree means very satisfied and strongly disagree is very unsatisfied.
To compare the time to initiating treatment after completing in-clinic versus at-home testing. | Six months after being consented to the study.
  The time to treatment initiation will be identified by the provider.

CONTACTS AND LOCATIONS:
Overall Officials: Yanett Anaya, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradshaw A, Ballon-Landa E, Owusu R, Hsieh TC. Poor Compliance With Postvasectomy Semen Testing: Analysis of Factors and Barriers. Urology. 2020 Feb;136:146-151. doi: 10.1016/j.urology.2019.10.026. Epub 2019 Nov 26. PMID 31778681
- [Background] Practice Committee of the American Society for Reproductive Medicine. Diagnostic evaluation of the infertile male: a committee opinion. Fertil Steril. 2015 Mar;103(3):e18-25. doi: 10.1016/j.fertnstert.2014.12.103. Epub 2015 Jan 15. PMID 25597249
- [Background] Infertility Workup for the Women's Health Specialist: ACOG Committee Opinion, Number 781. Obstet Gynecol. 2019 Jun;133(6):e377-e384. doi: 10.1097/AOG.0000000000003271. PMID 31135764
- [Background] Ethics Committee of the American Society for Reproductive Medicine. Disparities in access to effective treatment for infertility in the United States: an Ethics Committee opinion. Fertil Steril. 2015 Nov;104(5):1104-10. doi: 10.1016/j.fertnstert.2015.07.1139. Epub 2015 Sep 10. PMID 26364838
- [Background] Herndon CN, Anaya Y, Noel M, Cakmak H, Cedars MI. Outcomes from a university-based low-cost in vitro fertilization program providing access to care for a low-resource socioculturally diverse urban community. Fertil Steril. 2017 Oct;108(4):642-649.e4. doi: 10.1016/j.fertnstert.2017.06.035. Epub 2017 Sep 2. PMID 28874259